CLINICAL TRIAL: NCT05063188
Title: Is Connective Tissue Massage Effective In Individuals With Fibromyalgia?
Brief Title: Connective Tissue Massage With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Bilge Basakci Calik, Assoc. Prof., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Connective Tissue Massage
Record Dates: First submitted 2021-09-22; First posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Other: clinical pilates exercises
- Intervention group (Experimental)
  Interventions: Other: Connective Tissue Massage; Other: clinical pilates exercises

INTERVENTIONS:
Other: Connective Tissue Massage — Connective tissue massage was started from lumbosacral region and continued lower thoracic, scapular, interscapular, and cervical regions, respectively.
  Arms: Intervention group
Other: clinical pilates exercises — Exercises were applied 3 times for 6 weeks, a total of 18 sessions. One session consisted of 10 minutes of warm-up, 40 minutes of Clinical Pilates exercises and 10 minutes of cooling down (60 minutes in total).

SUMMARY:
The aim of the study was to examine the effectiveness of clinical pilates exercises and connective tissue massage in individuals with Fibromyalgia (FM). 32 women were randomly divided into two groups as intervention (n=15, mean age=48.80±7.48) and control (n=17, mean age=55.64±7.87). While connective tissue massage and clinical pilates exercises were applied to the intervention group, control group were applied only clinical pilates exercises.According to our results, connective tissue massage increased the effectiveness of clinical pilates exercises in individuals with FM.

ELIGIBILITY:
Inclusion Criteria:(a) having FM diagnosis according to American College of Rheumatology 2016 criteria, (b) being a women, (c) aged 20-65. (d) being stable in drug use for at least 6 months or more. (e) being volunteer to participate in this study.

-

Exclusion Criteria:(a) have been exercising regularly for the past three months, (b) the presence of uncontrolled cardiopulmonary disease, (c) the presence of orthopedic, neurological or mental problems that may prevent exercise, (d) having undergone any surgery in the last six months for both groups, (e) pregnancy, (f) presence of malignancy, (g) not being able to participate in at least 75% of the training.

-

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Pain Location Inventory | 10 min
Fibromyalgia Impact Questionnaire | 15 min
Health Assessment Questionnaire | 10 min
Beck Anxiety Inventory | 10 min
Short Form-36 | 10 min
Biopsychosocial Questionnaire | 15 min

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Pamukkale, Denizli, Turkey (Türkiye)